CLINICAL TRIAL: NCT04180345
Title: Flare_IBD: Development and Validation of a Questionnaire Based on Patients' Messages on an Internet Forum for Early Detection of Flare in Inflammatory Bowel Disease
Brief Title: Development of a Questionnaire Based on Patients' Messages on an Internet Forum for Flare Detection in IBD
Acronym: FLARE_IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Association François Aupetit, Paris, France (Unknown); University of Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01520-57
Record Dates: First submitted 2019-10-23; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Flare; Inflammatory Bowel Diseases; Questionnaire; Internet; Mixed methods
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validation of the questionnaire: Items reduction, ajustment and psychometric validation of the questionnaire
  Interventions: Other: Psychometric validation of the questionnaire

INTERVENTIONS:
Other: Psychometric validation of the questionnaire — Delph Process : expert panel will include HCPs and patients. They will evaluate the relevance of items on a Likert scale (HCPs N = 25 ; Patients N = 25 ) "Think aloud" interviews (N = 10 patients) Psychometric validation ( N = 200 patients)

SUMMARY:
Crohn's disease and ulcerative colitis, the two major forms of inflammatory bowel disease (IBD) are chronic disabling conditions characterized by flares followed by periods of remission. However, IBD patients are seen every 3 to 6 months in the outpatient clinic, and the occurrence of a flare between two outpatient visits is not captured. In the current state of knowledge, there is no validated patient-reported outcome (PRO) tool to measure the phenomenon of flare in IBD. This study aimed to use an innovative methodology to collect messages posted by patients in an Internet forum for developing and validating a PRO measuring flare in IBD.

The design involves 1) Engineering sciences for scraping extraction of messages posted in an Internet forum and for Identification of messages related to flare, 2) Qualitative methods for thematic content analyze of the messages posted, for candidate items generation, for items selection (Delphi process) and for items adjustment ("think aloud" interviews), 3) Quantitative methods for psychometric validation of the PRO.

ELIGIBILITY:
Inclusion Criteria:

* Every patient consulting the gastroenterology unit of Nancy University Hospital with a confirmed IBD diagnosis, regardless of the patient's state or treatment will be considered for inclusion

Exclusion Criteria:

* patients with a diagnosis < 3 months.
* Protected persons (minors, adults under guardianship, pregnant or breastfeeding women, people living in a public health or social institution, patients in an emergency situation, incarcerated individuals)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crohn's disease and ulcerative colitis, the two major forms of inflammatory bowel disease are chronic disabling conditions characterized by flares followed by periods of remission. To the current state of knowledge, there is no validated patient-reported outcome (PRO) tool to measure the phenomenon of flare in inflammatory bowel disease. This study aimed to use an innovative methodology to collect messages posted by patients in an Internet forum for developing and validating a PRO measuring flare in inflammatory bowel disease.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Scale calibration of the new developped questionnaire | About 30 minutes
  Weighing scale calibration
Construct validity of the new developped questionnaire | About 30 minutes
  Exploratory factor analysis, discriminant validity by Kruskal-Wallis tests
Convergence proprieties of the new developped questionnaire | about 30 minutes
  Convergence test of Flare-IBD scores with objective biological markers and clinical markers used in routine clinical practice
Reproductibility of the new developped questionnaire | Up to 8 days
  Investigation of test-retest reliability with a second questionnaire administered 8 days later.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ricci L, Epstein J, Buisson A, Devos C, Toussaint Y, Peyrin-Biroulet L, Guillemin F. Flare-IBD: development and validation of a questionnaire based on patients' messages on an internet forum for early detection of flare in inflammatory bowel disease: study protocol. BMJ Open. 2020 Jul 1;10(7):e037211. doi: 10.1136/bmjopen-2020-037211. PMID 32611745